CLINICAL TRIAL: NCT05881603
Title: Prevalence of Venous conGestion and Its Association With Renal Injuries Evaluated by the VExUS Score On Admission With UltraSound in Patients With Cardiogenic Pulmonary Edema
Acronym: GRIEVOUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/CHU/22; 2022-A02815-38 (Other: id-RCB)
Record Dates: First submitted 2023-05-05; First posted 2023-05-31 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cardiogenic Acute Pulmonary Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: " VExUS score " (Venous Excess Ultrasound Score) — " VExUS score " (Venous Excess Ultrasound Score)

SUMMARY:
Acute respiratory distress (ARD) is a frequent reason for seeking care in emergency medicine and represents an important cause of morbidity and mortality. Among the various etiologies, Acute Cardiogenic Pulmonary Edema (C APE) currently represents one of the main causes of ARD, particularly in the elderly, with a prevalence of 43% and an estimated mortality of 21%. According to the recommendations issued in 2021 by the European Society of Cardiology (ESC), the treatment of cardiogenic APE is currently based on a triptych combining:

* Oxygen therapy with an Saturation of Hemoglobin with Oxygen (SpO2) target > 94% and the use of non-invasive ventilation (NIV),
* A vasodilator administered intravenously (IV),
* A loop diuretic by IV route. Although most C APE are today considered to occur in a context of hypervolaemia and are uniformly treated by the administration of diuretics according to the recommendations in force, several works underline the fact that a non-negligible part of these clinical pictures would occur in patients with no water and sodium overload but with "relative" hypervolaemia masking euvolaemia or even hypovolaemia.

At present, no additional examination is recommended to determine the patient's volume status. However, it has been shown more recently that some patients who do not have absolute hypervolaemia could develop acute renal complications during treatment for C APE. In addition, systematic treatment with loop diuretics in patients without absolute hypervolaemia could be harmful by inducing post-treatment hypovolaemia.

At the present time, there are no data from the literature having been interested in the possible association existing between the state of blood volume of the patient on admission and the occurrence of renal complications in the aftermath of the treatment. initial. The prevalence of renal complications was nevertheless evaluated at 9% in this category of patients. The estimated prevalence of this complication and its particular seriousness, particularly in the case of chronic acute kidney injury, as well as its cost to society, justify carrying out a study aimed at evaluating the prevalence of venous congestion in the acute phase and of its possible association with the occurrence of renal complications in the course of this.

Among the various methods for assessing blood volume status, there is a growing literature regarding the use of clinical ultrasound in emergency medicine (ECMU). More recently, an ultrasound score called "VExUS score" (Venous Excess Ultrasound Score) has been developed. This offers the possibility of evaluating and classifying in 4 grades of increasing severity, simply and quickly, the state of venous congestion of patients. This score is based on the presence or absence of venous Doppler ultrasound abnormalities assessed at the level of the inferior vena cava, at the level of the supra-hepatic veins, of the portal and renal venous flow. This score, adapted to the practice of ECMU and making it possible to distinguish patients with or without venous congestion criteria, could provide arguments to guide diuretic treatment by offering personalized care. This evaluation would ultimately make it possible to offer diuretic treatment only in the event of signs suggestive of absolute hypervolaemia and thus avoid the occurrence of complications related to inappropriate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of cardiogenic Acute Pulmonary Edema defined by the association of clinical acute respiratory distress (current breath rate > 25/min, indrawing, flapping of the wings of the nose, thoraco-abdominal rocking, signs of hypoxemia, signs of hypercapnia) AND signs of pulmonary overload (clinical, biological and radiological arguments).
* Having given their non-objection to participation in the study (or non-objection of a loved one in an emergency context)

Exclusion Criteria:

* Breastfeeding in progress
* Known hypersensitivity to furosemide
* History of kidney transplantation
* Known water and electrolyte disorder
* Hepatic encephalopathy
* Suspicion of obstruction in the urinary tract
* Person deprived of liberty by judicial or administrative decision, minor, person subject to a measure of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cardiogenic Acute Pulmonary Edema
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Estimate the prevalence of the different grades of venous congestion assessed by the VExUS score in ultrasound | within 12 hours of admission
  VExUS score in ultrasound score 0 to 3 / Higher score means worse outcome

SECONDARY OUTCOMES:
Evaluate the association between the different ultrasound grades of venous congestion described by the ultrasound VExUS score and the occurrence of renal complications during hospitalization defined by the MAKE-Discharge | 7 days, 30 days, 180 days
  Major Adverse Kidney Events (MAKE), composite criterion :
  - Criterion 1 : De novo acute renal failure (ARI) or worsening of pre-existing chronic renal failure (CRI), defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) reference classification
Evaluate the association between the different ultrasound grades of venous congestion described by the ultrasound VExUS score and the occurrence of renal complications during hospitalization defined by the MAKE-Discharge | 7 days, 30 days, 180 days
  Major Adverse Kidney Events (MAKE), composite criterion :
  * Criterion 2 : Need for de novo extra-renal purification (ERT) or increased frequency of use of ERT or need for emergency ERT in a patient usually on dialysis,
  * Occurrence of a death.
Evaluate the association between the different ultrasound grades of venous congestion described by the ultrasound VExUS score and the occurrence of renal complications during hospitalization defined by the MAKE-Discharge | 7 days, 30 days, 180 days
  Major Adverse Kidney Events (MAKE), composite criterion :
  * Criterion 3 : Occurence of death
  * Occurrence of a death.
Assess the association between the grade of the VExUS ultrasound score on admission and the total and daily dose of furosemide administered to the patient | 7 days
  dose of furosemide
Evaluate the kinetics of evolution of the VExUS ultrasound score performed at the patient's bedside in comparison with the values found on admission | within 12 hours of admission , day 3 day 7
  VExUS score in ultrasound score 0 to 3 / Higher score means worse outcome
Evaluate the association between the presence of venous congestion (VExUS score ≥ 1) or not and vital and functional status : Gerontological autonomy iso-resource groups | day 7, day 30, day 180
  Gerontological autonomy iso-resource groups (score AGGIR) Value 1 to 6 / Higher score mean better outcome
Evaluate the association between the presence of venous congestion (VExUS score ≥ 1) or not and vital and functional status : Activities of daily living | day 7, day 30, day 180
  Activities of daily living (score ADL) Value 1 to 6 / Higher score mean better outcome
Evaluate the association between the presence of venous congestion (VExUS score ≥ 1) or not and vital and functional status : Barthel Index | day 7, day 30, day 180
  Barthel Index Value 0 to 100 / Higher score mean better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Denis, France